CLINICAL TRIAL: NCT00591383
Title: Phase I Study of Indibulin in Combination With Erlotinib in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBL1004
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Solid Tumors
Keywords: Cancer; Indibulin; Erlotinib
MeSH Terms: conditions — Neoplasms | interventions — indibulin; Erlotinib Hydrochloride

ARMS (1):
- Single Arm (Experimental): Once Maximum Tolerated Dose (MTD) is determined an expanded cohort will be enrolled to evaluate efficacy.
  Interventions: Drug: indibulin; Drug: erlotinib

INTERVENTIONS:
Drug: indibulin — indibulin, dose escalation, 200 mg - 600 mg. Taken twice every day.
  Other Names: ZIO-301
Drug: erlotinib — erlotinib taken at 150 mg every morning with food.

SUMMARY:
Single arm, open label, Phase I, dose-escalation study of indibulin in combination with erlotinib in subjects with advanced histologically confirmed, solid tumors for which no standard therapy exists and for whom treatment with erlotinib is considered medically acceptable.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with advanced, histologically confirmed solid tumors for which no standard therapy exists and for whom treatment with erlotinib is considered medically acceptable.
2. ≥18 years of age
3. ECOG performance score ≤2
4. Eligible subjects MUST have at least one measurable lesion as defined by RECIST guidelines. Measurable lesions MUST NOT have been in a previously irradiated field or injected with biological agents.
5. Life-expectancy ≥12 weeks
6. No more than 2 prior chemotherapy regimens for metastatic disease
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted <2 weeks prior to Study Day 1:

   * Creatinine ≤1.5×upper limit of normal (ULN) OR a calculated creatinine clearance ≥50 cc/min
   * Total bilirubin ≤1.5×ULN
   * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤2.5×ULN
   * White blood cell count ≥3.0×109/L
   * Absolute Neutrophil Count (ANC) ≥1.5×109/L
   * Platelets ≥100×109/L
   * Hemoglobin ≥10 g/dL
8. Written informed consent in compliance with ZIOPHARM policies and the Human Investigation Review Committee with jurisdiction over the site.
9. Each man and woman of childbearing potential must agree to use a reliable method of contraception during the study and for 3 months following the last dose of study drug.

Exclusion Criteria:

1. New York Heart Association (NYHA) functional class ≥3 or myocardial infarction within 6 months (see Appendix 5)
2. Uncontrolled cardiac arrhythmia other than asymptomatic atrial fibrillation
3. Subjects cannot be receiving cytochrome P450-inducing anticonvulsants (EIAEDs: eg, phenytoin, carbamazepine, phenobarbital, primidone, oxcarbezine)
4. Subjects may not be taking CYP3A4 inducers (rifampicin)
5. Subjects must not have any evidence of bleeding diathesis or coagulopathy
6. Subjects with international normalized ration (INR) >1.5 are excluded, unless the subject is on full dose warfarin
7. Subjects on full-dose anticoagulants (eg, warfarin) are eligible provided that both of the following criteria are met:

   * The subject has an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
   * The subject has no active bleeding or pathological condition that carries a high risk of bleeding (eg, tumor involving major vessels or known varices.
8. Subjects on prophylactic anticoagulation (ie, low-dose warfarin) are eligible provided their coagulation parameter levels are as follows: prothrombin time (INR of prothrombin time) <1.1×institutional ULN
9. Pregnancy and/or lactation
10. Uncontrolled systemic infection (documented with microbiological studies)
11. Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry. Mitomycin C or nitrosureas should not be given within 6 weeks of study entry.
12. Prior treatment with EGFR inhibitors
13. Radiotherapy during the study or within 3 weeks of study entry
14. Surgery within 4 weeks of start of study drug excluding tumor biopsy for pharmacodynamic parameters
15. Investigational drug therapy outside of this trial during or within 4 weeks of study entry
16. History of an invasive second primary malignancy diagnosed within the previous 3 years except for Stage I endometrial/cervical carcinoma or prostate carcinoma treated surgically, and non-melanoma skin cancer
17. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
18. Any condition that is unstable or could jeopardize the safety of the subject and his/her compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
toxicities | 6 months

SECONDARY OUTCOMES:
pharmacokinetics | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lewis, MD, Study Director — Alaunos Therapeutics
Locations (1):
- Houston, Texas, United States

REFERENCES:
- [Derived] Kapoor S, Srivastava S, Panda D. Indibulin dampens microtubule dynamics and produces synergistic antiproliferative effect with vinblastine in MCF-7 cells: Implications in cancer chemotherapy. Sci Rep. 2018 Aug 17;8(1):12363. doi: 10.1038/s41598-018-30376-y. PMID 30120268